CLINICAL TRIAL: NCT05881005
Title: Prévalence De La Stéato-fibrose Hépatique Dans Le Syndrome De Cushing
Brief Title: NAC- NAFLD and Cushing
Acronym: NAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC22-0389; 2023-A00727-38 (Other: ANSM)
Record Dates: First submitted 2023-05-05; First posted 2023-05-30 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Cushing Syndrome; Fatty Liver Disease
MeSH Terms: conditions — Cushing Syndrome; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- open-label study (Other): hepatic MRI, Fibroscan
  Interventions: Diagnostic Test: hepatic MRI

INTERVENTIONS:
Diagnostic Test: hepatic MRI — Quantification of hepatic steatosis with RMI at the diagnosis (T0) and one year after remission (T1). The percentage of patients with complete resolution of hepatic steatosis on MRI will be determined.
  Other Names: Fibroscan

SUMMARY:
Cushing's Syndrome is a rare disease resulting from prolonged exposure to high levels of circulating cortisol. Clinical manifestations are variable but many patients present a metabolic syndrome (abdominal obesity, insulin resistance, dyslipidemia, hypertension). With regard to the liver, experimental data have shown that excess cortisol leads in an increase in lipogenesis and a reduction in the oxidation of fatty acids. This, in association with an accumulation of visceral adipose tissue and deregulation of adipokines, may contribute to the development of hepatic steatosis in animals. However, few data is available in humans with only one study of 50 patients with Cushing's syndrome estimating the prevalence of hepatic steatosis at 20%.

NAFLD (Non-Alcoholic Fatty Liver Disease), is defined as the presence of hepatic steatosis in the absence of secondary causes of intrahepatic fat accumulation. It is a heterogeneous disease ranging from simple liver steatosis, whose prognosis is generally considered to be benign, to inflammation (NASH, Non-Alcoholic Steato-Hepatitis) which may progress to fibrosis, cirrhosis and an increased risk of hepatocellular carcinoma. The prognosis for NAFLD is mainly related to the severity of hepatic fibrosis.

In Cushing's syndrome, normalization of cortisol production is the most effective strategy to improve co-morbidities associated with hypercortisolism. However, some of these complications, especially the metabolic co morbidities, could not be completely reversible and no data is available about resolution of hepatic steatosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Active Cushing's syndrome

Exclusion Criteria:

* Other common causes of chronic liver disease (HBV, HCV, haemochromatosis, alcohol)
* Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-10-28 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
Frequency of resolution of hepatic steatosis | 2 years
  To evaluate the frequency of complete resolution of hepatic steatosis in patients with cushing syndrome after remission of hypercortisolism

SECONDARY OUTCOMES:
Prevalence of steatosis at diagnosis of Cushing | 2 years
  to assess the prevalence of hepatic steatosis at the diagnosis of Cushing's syndrome.
Prevalence of steatosis at diagnosis of Cushing | 2 years
  to evaluate the prevalence of steatosis
Fatty Liver Index (non-invasive biomarkers of hepatic steatosis ) | 2 years
  to evaluate the non-invasive biomarkers of hepatic steatosis (Fatty Liver Index)
FIB-4 (non-invasive biomarkers advanced hepatic fibrosis) | 2 years
  to evaluate the non-invasive biomarkers advanced hepatic fibrosis (FIB-4)
e-LIFT (non-invasive biomarkers advanced hepatic fibrosis) | 2 years
  to evaluate the non-invasive biomarkers advanced hepatic fibrosis ( e-LIFT, NAFLD Fibrosis Score)
NAFLD Fibrosis Score (non-invasive biomarkers advanced hepatic fibrosis) | 2 years
  to evaluate the non-invasive biomarkers advanced hepatic fibrosis (NAFLD Fibrosis Score)
Prevalence of steatosis at diagnosis of Cushing | 2 years
  4. To assess the performance of CAP (Controlled Attenuation Parameter) in the diagnosis of hepatic steatosis in Cushing's syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Claire BRIET, Principal Investigator — University Hospital of Anger
Locations (6):
- France (6):
  - University Hospital, Angers, Angers
  - University Hospital, Bordeaux, Bordeaux
  - University Hospital, Brest, Brest
  - University Hospital, Grenoble, Grenoble
  - University Hospital, Nantes, Nantes
  - University Hospital, Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No